CLINICAL TRIAL: NCT00464672
Title: A Phase III, Observer-Blind, Randomized, Controlled, Multicenter Study to Evaluate Safety, Tolerability, and Immunogenicity of Two Trivalent Subunit Inactivated Influenza Vaccines in Healthy Children Aged 3 to 8 Years, in Healthy Children/Adolescents Aged 9 to 17 Years,and in Healthy Adults Aged 18 to 64 Years
Brief Title: Safety, and Immunogenicity of Two Influenza Vaccines in Healthy Subjects 3 to 64 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Novartis Vaccines and Diagnostics, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V71P5; IND: 13299
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Results first posted 2010-05-05 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Influenza
Keywords: Influenza, Egg-Derived, Healthy Children, Healthy Adolescents, Healthy Adults, Safety, Immunogenicity, Trivalent, Inactivated, Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza virus vaccine (Experimental)
  Interventions: Biological: Influenza virus vaccine
- Comparator influenza vaccine (Active Comparator)
  Interventions: Biological: Comparator influenza vaccine

INTERVENTIONS:
Biological: Influenza virus vaccine — Two intramuscular injections of the investigational influenza virus vaccine administered 4 weeks part to group 3 to 8 years of age while one injection was administered to groups 9 to 17 years of age and 18 to 64 years of age.
  Arms: Influenza virus vaccine
Biological: Comparator influenza vaccine — Two intramuscular injections were administered 4 weeks apart to group 3 to 8 years of age while one injection was administered to groups 9 to 17 years of age and 18 to 64 years of age.
  Arms: Comparator influenza vaccine

SUMMARY:
This protocol is designed to evaluate safety, clinical tolerability and immunogenicity of the 2007 southern hemisphere formulation of a Novartis conventional influenza vaccine licensed in the EU and many other worldwide countries, according to the US FDA Draft Guidance for Industry "Clinical data needed to support the licensure of trivalent inactivated influenza vaccine", issued in March 2006, and to evaluate safety, clinical tolerability and immunogenicity of the 2007 southern hemisphere formulation of a Novartis conventional influenza vaccine already licensed in US. The purpose of the control arm is primarily to provide a comparative assessment for safety, not immunogenicity or effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects 3 to 64 years of age

Exclusion Criteria:

* Receipt of other investigational products within 3 months or other vacine within 1 month;
* Allergy to eggs, egg products, or any other vaccine component;
* Laboratory confirmed influenza disease within 6 months;
* Have previously received an influenza vaccination (3 to 8 years only);

Ages: 3 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1893 (Actual)
Dates: Start 2007-04; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Director — Novartis
Locations (2):
- Argentina (2):
  - Site 2: C1425AWK, Buenos Aires
  - Site 1: X5000BJH, Córdoba

REFERENCES:
- [Derived] Tregnaghi MW, Stamboulian D, Vanadia PC, Tregnaghi JP, Calvari M, Fragapane E, Casula D, Pellegrini M, Groth N. Immunogenicity, safety, and tolerability of two trivalent subunit inactivated influenza vaccines: a phase III, observer-blind, randomized, controlled multicenter study. Viral Immunol. 2012 Jun;25(3):216-25. doi: 10.1089/vim.2011.0063. PMID 22691101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 6 weeks for enrollment with date of first enrolment on April 2007
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- Influenza Virus Vaccine (18 to 64 Years); Influenza Virus Vaccine (9 to 17 Years): One injection of the investigational influenza virus vaccine was administered intramuscularly
- Comparator Influenza Vaccine (18 to 64 Years); Comparator Influenza Vaccine (9 to 17 Years): One injection of the comparator influenza vaccine was administered intramuscularly
- Influenza Virus Vaccine (3 to 8 Years): Two injections of the investigational influenza virus vaccine were administered intramuscularly
- Comparator Influenza Vaccine (3 to 8 Years): Two injections of the comparator influenza vaccine were administered intramuscularly
Period: Overall Study
Arm/Group | Influenza Virus Vaccine (18 to 64 Years) | Comparator Influenza Vaccine (18 to 64 Years) | Influenza Virus Vaccine (9 to 17 Years) | Comparator Influenza Vaccine (9 to 17 Years) | Influenza Virus Vaccine (3 to 8 Years) | Comparator Influenza Vaccine (3 to 8 Years)
Started | 460 | 232 | 400 | 200 | 402 | 199
Completed | 435 | 222 | 400 | 199 | 392 | 195
Not Completed | 25 | 10 | 0 | 1 | 10 | 4
Not completed — withdrawal of consent | 0 | 0 | 0 | 1 | 9 | 4
Not completed — Lost to Follow-up | 25 | 10 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Influenza Virus Vaccine: Injections of the investigational influenza virus vaccine were administered intramuscularly
- Comparator Influenza Vaccine: Injections of the comparator influenza vaccine were administered intramuscularly
- Total: Total of all reporting groups
Arm/Group | Influenza Virus Vaccine | Comparator Influenza Vaccine | Total
Number analyzed (Participants) | 1262 | 631 | 1893
Age, Continuous [Mean (Standard Deviation); unit: years]
  Chilren 3 to 8 years of age | 5.5 (1.7) | 5.4 (1.7) | 5.5 (1.7)
  Children/Adolescents 9 to 17 years of age | 12.7 (2.6) | 12.8 (2.6) | 12.7 (2.6)
  Adults 18 to 64 years of age | 38.8 (14.4) | 37.8 (12.6) | 38.5 (12.5)
Sex/Gender, Customized [Number; unit: participants]
  Male | 575 | 294 | 869
  Female | 687 | 337 | 1024
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1168 | 579 | 1747
  Hispanic | 92 | 52 | 144
  Asian | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Seroprotection, in Healthy Adults 18 to 64 Years of Age
Description: To evaluate immunogenicity, measured by seroprotection (percentage of subjects achieving a hemagglutination inhibition [HI] titer ≥40) after one injection of the investigational influenza virus vaccine, administered to healthy adults 18 to 64 years of age. The CBER Guidance states that the lower bound of the two-sided 95% CI for the percentage of subjects achieving seroprotection meet or exceed 70%.
Time Frame: 21 days after vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Mean (95% Confidence Interval); unit: Percentages of participants
Groups:
- Influenza Virus Vaccine (A/H1N1); Influenza Virus Vaccine (A/H3N2); Influenza Virus Vaccine (Strain B): One injection of the investigational influenza virus vaccine was administered intramuscularly
- Comparator Influenza Vaccine (A/H1N1); Comparator Influenza Vaccine (A/H3N2); Comparator Influenza Vaccine (Strain B): One injection of the comparator influenza vaccine was administered intramuscularly
Arm/Group | Influenza Virus Vaccine (A/H1N1) | Influenza Virus Vaccine (A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (A/H1N1) | Comparator Influenza Vaccine (A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 424 | 424 | 424 | 219 | 219 | 219
Percentages of participants | 93 [90 to 95] | 96 [94 to 98] | 91 [87 to 93] | 99 [97 to 100] | 100 [98 to 100] | 86 [81 to 91]

2. Primary Outcome: Percentage of Subjects Achieving a Seroconversion Rate, in Adults 18 to 64 Years of Age
Description: Seroconversion rate is defined as percentage of subjects achieving seroconversion (defined as negative pre-vaccination serum [HI<10]/ post-vaccination HI titer ≥40) or significant increase defined as at least a 4-fold increase). According to the CBER Guidance, the lower bound of the two-sided 95% CI for the percentage of subjects achieving seroconverion/significant increase meet or exceed 40%.
Time Frame: 21 days after vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Influenza Virus Vaccine (A/H1N1) | Influenza Virus Vaccine (A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (A/H1N1) | Comparator Influenza Vaccine (A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 424 | 424 | 424 | 219 | 219 | 219
Percentage of participants | 74 [69 to 78] | 72 [68 to 76] | 77 [72 to 81] | 86 [81 to 90] | 89 [84 to 92] | 74 [68 to 80]

3. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Symptoms in Adults 18 to 64 Years of Age
Description: Solicited local and systemic reactions were assessed after vaccination in adults 18 to 64 years of age.
Time Frame: 7 days after vaccination
Population: The analysis was performed on the safety population.
Measure: Number; unit: participants
Groups:
- Influenza Virus Vaccine: One injection of the investigational influenza virus vaccine was administered intramuscularly
- Comparator Influenza Vaccine: One injection of the comparator influenza vaccine was administered intramuscularly
Arm/Group | Influenza Virus Vaccine | Comparator Influenza Vaccine
Number analyzed (Participants) | 460 | 233
participants
  Any local reaction | 161 | 89
  Erythema | 27 | 12
  Induration | 38 | 24
  Swelling | 29 | 15
  Ecchymosis | 24 | 15
  Pain | 117 | 70
  Any Systemic Reaction | 147 | 84
  Chills | 21 | 17
  Malaise | 55 | 27
  Myalgia | 66 | 37
  Arthralgia | 30 | 14
  Headache | 108 | 42
  Sweating | 24 | 11
  Fatigue | 46 | 24
  Fever | 10 | 6

4. Secondary Outcome: Percentage of Subjects With Seroprotection, in Healthy Children/Adolescents 9 to 17 Years of Age
Description: To descriptively evaluate immunogenicity, measured by seroprotection rate (percentage of subjects achieving a hemagglutination inhibition [HI] titer ≥40) after one injection of investigational influenza virus vaccine, administered to healthy children/adolescents 9 to 17 years of age.
Time Frame: 21 days after vaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Mean (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Influenza Virus Vaccine (A/H1N1) | Influenza Virus Vaccine (A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (A/H1N1) | Comparator Influenza Vaccine (A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 393 | 393 | 393 | 192 | 192 | 192
Percentage of subjects | 99 [97 to 100] | 100 [99 to 100] | 93 [90 to 95] | 98 [96 to 100] | 100 [98 to 100] | 89 [84 to 93]

5. Secondary Outcome: Percentage of Subjects Achieving Seroconversion Rate, in Healthy Children/Adolescents 9 to 17 Years of Age
Description: Seroconversion rate is defined as percentage of subjects achieving seroconversion (defined as negative pre-vaccination serum [HI<10]/ post-vaccination HI titer ≥40) or significant increase (defined as at least a 4-fold increase) after one injection of the investigational influenza virus vaccine, administered to healthy children/adolescents 9 to 17 years of age.
Time Frame: 21 days after vaccination
Population: The analysis was performed on the per-protocol (PP)population.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Influenza Virus Vaccine (A/H1N1) | Influenza Virus Vaccine (A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (A/H1N1) | Comparator Influenza Vaccine (A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 393 | 393 | 393 | 192 | 192 | 192
Percentage of participants | 92 [88 to 94] | 67 [62 to 72] | 81 [76 to 84] | 91 [86 to 94] | 92 [87 to 95] | 73 [67 to 80]

6. Secondary Outcome: Geometric Mean Titers (GMTs), in Healthy Children/Adolescents 9 to 17 Years of Age
Description: To evaluate immunogenicity measured by GMTs after one injection of investigational influenza virus vaccine, administered to healthy children/adolescents 9 to 17 years of age.
Time Frame: 21 days after vaccination
Population: The analysis was performed on the per-protocol (PP)population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influenza Virus Vaccine (A/H1N1) | Influenza Virus Vaccine (A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (A/H1N1) | Comparator Influenza Vaccine (A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 393 | 393 | 393 | 192 | 192 | 192
Titers | 960 [857 to 1076] | 493 [453 to 536] | 144 [127 to 163] | 1246 [1058 to 1467] | 1463 [1296 to 1651] | 114 [95 to 136]

7. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Symptoms in Children/Adolescents 9 to 17 Years of Age
Description: Solicited local and systemic reactions were assessed after vaccination in children/adolescents 9 to 17 years of age.
Time Frame: 7 days after vaccination
Population: The analysis was performed on the safety population.
Measure: Number; unit: Participants
Groups:
- Influenza Virus Vaccine: Injection of the investigational influenza virus vaccine were administered intramuscularly
- Comparator Influenza Vaccine: Injection of the comparator influenza vaccine were administered intramuscularly
Arm/Group | Influenza Virus Vaccine | Comparator Influenza Vaccine
Number analyzed (Participants) | 400 | 199
Participants
  Any local reaction | 134 | 62
  Erythema | 7 | 3
  Induration | 28 | 13
  Swelling | 28 | 14
  Ecchymosis | 9 | 1
  Pain | 117 | 58
  Any Systemic reaction | 91 | 49
  Chills | 18 | 11
  Malaise | 18 | 8
  Myalgia | 35 | 25
  Arthralgia | 11 | 5
  Headache | 52 | 22
  Sweating | 4 | 3
  Fatigue | 25 | 9
  Fever | 1 | 4

8. Secondary Outcome: Percentage of Subjects With Seroprotection, in Healthy Children 3 to 8 Years of Age
Description: To descriptively evaluate immunogenicity, measured by seroprotection rate (percentage of subjects achieving a hemagglutination inhibition [HI] titer ≥40) after two injections of the investigational influenza virus vaccine, in healthy children 3 to 8 years of age.
Time Frame: 50 days after last vaccination
Population: The analysis was performed on the per-protocol (PP) population
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Groups:
- Influenza Virus Vaccine (A/H1N1); Influenza Virus Vaccine (A/H3N2); Influenza Virus Vaccine (Strain B): Two injections of the investigational influenza virus vaccine were administered intramuscularly
- Comparator Influenza Vaccine (A/H1N1); Comparator Influenza Vaccine (A/H3N2); Comparator Influenza Vaccine (Strain B): Two injections of the comparator influenza vaccine were administered intramuscularly
Arm/Group | Influenza Virus Vaccine (A/H1N1) | Influenza Virus Vaccine (A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (A/H1N1) | Comparator Influenza Vaccine (A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 296 | 296 | 296 | 149 | 149 | 149
Percentage of participants | 97 [94 to 99] | 100 [99 to 100] | 85 [80 to 89] | 99 [95 to 100] | 99 [96 to 100] | 81 [73 to 87]

9. Secondary Outcome: Percentage of Subjects Achieving Seroconversion Rate, in Healthy Children 3 to 8 Years of Age
Description: Seroconversion rate is defined as percentage of subjects achieving seroconversion (defined as negative pre-vaccination serum [HI<10]/ post-vaccination HI titer ≥40) or significant increase (defined as at least a 4-fold increase) after two injections of the investigational influenza virus vaccine, in healthy children 3 to 8 years of age.
Time Frame: 50 days after last vaccination
Population: The analysis was performed on the per protocol (PP) population.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Influenza Virus Vaccine (A/H1N1) | Influenza Virus Vaccine (A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (A/H1N1) | Comparator Influenza Vaccine (A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 296 | 296 | 296 | 149 | 149 | 149
Percentage of participants | 95 [91 to 97] | 86 [82 to 90] | 83 [78 to 87] | 97 [92 to 99] | 95 [90 to 98] | 79 [72 to 85]

10. Secondary Outcome: Geometric Mean Titers (GMTs), in Healthy Children 3 to 8 Years of Age
Description: To evaluate immunogenicity measured by GMTs after two injections of the investigational influenza virus vaccine, in healthy children 3 to 8 years of age.
Time Frame: 50 days after last vaccination
Population: The analysis was performed on the per-protocol (PP)population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influenza Virus Vaccine (A/H1N1) | Influenza Virus Vaccine (A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (A/H1N1) | Comparator Influenza Vaccine (A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 296 | 296 | 296 | 149 | 149 | 149
Titers | 625 [532 to 734] | 710 [637 to 792] | 157 [133 to 185] | 716 [570 to 898] | 1472 [1263 to 1715] | 126 [100 to 158]

11. Secondary Outcome: Number or Subjects Reporting Solicited Local and Systemic Symptoms, in Healthy Children 3 to 8 Years of Age.
Description: Solicited local and systemic reactions were assessed after each vaccination, in healthy children 3 to 8 years of age.
Time Frame: 7 days after each vaccination
Population: The analysis was performed on the safety population.
Measure: Number; unit: Participants
Groups:
- Influenza Virus Vaccine (Injection 1); Influenza Virus Vaccine (Injection 2): Injections of the investigational influenza virus vaccine were administered intramuscularly.
- Comparator Influenza Vaccine (Injection 1); Comparator Influenza Vaccine (Injection 2): Injections of the comparator influenza vaccine were administered intramuscularly.
Arm/Group | Influenza Virus Vaccine (Injection 1) | Comparator Influenza Vaccine (Injection 1) | Influenza Virus Vaccine (Injection 2) | Comparator Influenza Vaccine (Injection 2)
Number analyzed (Participants) | 402 | 199 | 396 | 197
Participants
  Any Local Reaction | 92 | 56 | 66 | 39
  Erythema | 9 | 5 | 3 | 3
  Induration | 11 | 10 | 13 | 8
  Swelling | 22 | 16 | 13 | 8
  Ecchymosis | 18 | 9 | 10 | 5
  Pain | 68 | 40 | 57 | 35
  Any Systemic Reaction | 66 | 38 | 41 | 21
  Chills | 10 | 8 | 8 | 5
  Malaise | 21 | 12 | 19 | 7
  Myalgia | 19 | 9 | 19 | 10
  Arthralgia | 5 | 2 | 5 | 1
  Headache | 28 | 18 | 15 | 11
  Sweating | 5 | 3 | 3 | 1
  Fatigue | 18 | 9 | 10 | 4
  Fever | 12 | 3 | 10 | 5

12. Secondary Outcome: Geometric Mean Titers (GMTs), in Healthy Adults 18 to 64 Years of Age
Description: Immunogenicity measured by GMTs after one injection of the investigational influenza virus vaccine, in healthy adults 18 to 64 years of age.
Time Frame: 21 days after vaccination
Population: The analysis was done on the per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influenza Virus Vaccine (A/H1N1) | Influenza Virus Vaccine (A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (A/H1N1) | Comparator Influenza Vaccine (A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 424 | 424 | 424 | 219 | 219 | 219
Titers | 244 [214 to 278] | 219 [196 to 245] | 126 [113 to 140] | 512 [426 to 615] | 485 [415 to 567] | 104 [90 to 122]

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events were collected from 21 days after the last vaccination (up to day 53) to study termination (up to day 216). All serious adverse events were collected throughout the entire study period (up to day 216).
Description: One subject (18 years of age) in the comparator influenza vaccine group was enrolled in the adolescent age strata but was included in the adult age stratum for the safety analyses.
Arm/Group | Influenza Virus Vaccine (18 to 64 Years) | Comparator Influenza Vaccine (18 to 64 Years) | Influenza Virus Vaccine (9 to 17 Years) | Comparator Influenza Vaccine (9 to 17 Years) | Influenza Virus Vaccine (3 to 8 Years) | Comparator Influenza Vaccine (3 to 8 Years)
Serious Adverse Events (participants affected / at risk) | 6/460 | 2/233 | 4/400 | 0/199 | 3/402 | 3/199
Other Adverse Events (participants affected / at risk) | 235/460 | 128/233 | 167/400 | 80/199 | 153/402 | 91/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza Virus Vaccine (18 to 64 Years) (N=460) | Comparator Influenza Vaccine (18 to 64 Years) (N=233) | Influenza Virus Vaccine (9 to 17 Years) (N=400) | Comparator Influenza Vaccine (9 to 17 Years) (N=199) | Influenza Virus Vaccine (3 to 8 Years) (N=402) | Comparator Influenza Vaccine (3 to 8 Years) (N=199)
Visual acuity reduced transiently (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dysentery (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza Virus Vaccine (18 to 64 Years) (N=460) | Comparator Influenza Vaccine (18 to 64 Years) (N=233) | Influenza Virus Vaccine (9 to 17 Years) (N=400) | Comparator Influenza Vaccine (9 to 17 Years) (N=199) | Influenza Virus Vaccine (3 to 8 Years) (N=402) | Comparator Influenza Vaccine (3 to 8 Years) (N=199)
Chills (General disorders) | 22 (25) | 18 (20) | 18 (24) | 11 (11) | 18 (19) | 12 (14)
Fatigue (General disorders) | 47 (51) | 24 (26) | 25 (25) | 9 (9) | 26 (28) | 12 (14)
Injection Site Erythema (General disorders) | 27 (27) | 12 (12) | 7 (7) | 3 (3) | 12 (12) | 7 (8)
Injection Site Haemorrhage (General disorders) | 25 (25) | 15 (15) | 9 (9) | 1 (1) | 26 (28) | 13 (14)
Injection Site Induration (General disorders) | 38 (38) | 24 (24) | 28 (28) | 13 (13) | 23 (24) | 16 (18)
Injection Site Pain (General disorders) | 117 (121) | 70 (70) | 117 (120) | 58 (58) | 97 (129) | 59 (75)
Injection Site Swelling (General disorders) | 29 (29) | 15 (15) | 28 (28) | 14 (14) | 34 (37) | 20 (24)
Malaise (General disorders) | 56 (61) | 28 (29) | 18 (18) | 8 (8) | 37 (41) | 19 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (38) | 15 (16) | 11 (11) | 5 (5) | 10 (12) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 66 (74) | 38 (39) | 35 (36) | 25 (26) | 34 (41) | 17 (19)
Headache (Nervous system disorders) | 111 (133) | 45 (54) | 52 (56) | 23 (29) | 41 (46) | 26 (30)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 24 (26) | 11 (14) | 4 (4) | 3 (3) | 8 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less